CLINICAL TRIAL: NCT02442258
Title: Evaluation of the Pharmacokinetics and Safety of ABT-493 and ABT-530 in Subjects With Normal and Impaired Renal Function
Brief Title: Pharmacokinetics and Safety of ABT-493 and ABT-530 in Subjects With Normal and Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M13-600
Record Dates: First submitted 2015-05-11; First posted 2015-05-13 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-02

CONDITIONS: Renal Impairment
Keywords: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — glecaprevir; pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 - Mild Renal Impairment (Experimental): Subjects with mild renal impairment. eGFR (by MDRD equation) range 60 - 89 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group 2 - Moderate Renal Impairment (Experimental): Subjects with moderate renal impairment. eGFR (by MDRD equation) range 30 - 59 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group 3 - Severe Renal Impairment (Experimental): Subjects with severe renal impairment. eGFR (by MDRD equation) range 15 - 29 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group 4 - End Stage Renal Disease, Not Yet on Dialysis (Experimental): Subjects with end stage renal disease, not yet on dialysis. eGFR (by MDRD equation) range < 15 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group 5 - Normal Renal Function (Experimental): Subjects with normal renal function. eGFR (by MDRD equation) range ≥ 90 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530
- Group 6 - End Stage Renal Disease, Requiring Dialysis. (Experimental): Subjects with end stage renal disease, requiring dialysis. eGFR (by MDRD equation) < 15 mL/min/1.73 m2 as determined at Screening.
  Interventions: Drug: ABT-493; Drug: ABT-530

INTERVENTIONS:
Drug: ABT-493 — A single dose of ABT-493 will be given orally in combination with ABT-530.
Drug: ABT-530 — A single dose of ABT-530 will be given orally in combination with ABT-493.

SUMMARY:
This is an open-label, single dose study designed to assess the pharmacokinetics and safety of ABT-493 and ABT-530 in subjects with either normal renal function or impaired renal function.

DETAILED DESCRIPTION:
Up to 48 subjects will be selected and enrolled according to the subject selection criteria: 8 subjects with mild renal impairment (Group 1), 8 subjects with moderate renal impairment (Group 2), 8 subjects with severe renal impairment (Group 3), 8 subjects with end stage renal disease that are not yet on dialysis (Group 4), 8 healthy subjects with normal renal function (Group 5), and 8 subjects with end stage renal disease on hemodialysis (Group 6).

ELIGIBILITY:
Inclusion Criteria: All Subjects

* Females must have negative results for pregnancy tests performed:

  * At Screening on a urine specimen, and
  * On a serum sample obtained on Study Day -2 (prior to dosing).
* Body Mass Index (BMI) is ≥ 18 to ≤ 38 kg/m2, inclusive.
* Body Weight > 50 kg.

Subjects with Normal Renal Function

In addition to the main inclusion criteria above for all subjects, the following criteria must be met for subjects with normal renal function enrolled in Group 5:

* Judged to be in general good health based upon the results of a medical history, physical examination, and 12-lead electrocardiogram (ECG).
* At screening, estimated GFR (by MDRD equation) should be ≥ 90 mL/min/1.73 m2.

Subject with Renal Impairment

In addition to the main inclusion criteria for all subjects, the following criteria must be met for all subjects with renal impairment enrolled in Groups 1, 2, 3, 4 and 6:

* Judged to be in stable condition and acceptable for study participation based upon the results of a medical history, physical examination, laboratory profile and ECG.
* Presence of chronic renal impairment as indicated by medical history and a screening estimated GFR (by MDRD equation) < 90 mL/min/1.73 m2.
* Subjects with ESRD undergoing hemodialysis should have been receiving dialysis for at least 1 month.

Exclusion Criteria: - History of significant sensitivity to any drug.

* Pregnant or breastfeeding female.
* Recent (6-month) history of drug or alcohol abuse.
* Positive test result for hepatitis A virus immunoglobulin M (HAV-IgM), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or HIV antibodies (HIV Ab). Negative HIV status will be confirmed at Screening and the results will be maintained confidentially by the study site.
* Subjects on strict vegetarian diet.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
(SUB-STUDY 1) Area under the plasma concentration-time curve (AUC) from time 0 to infinity for the ABT-493 study drug. | Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1.
  The AUC from time 0 to infinity represents the total drug exposure over time.
Overall measurement of safety parameters | SUB-STUDY 1 - Duration of 14 days SUB-STUDY 2 - Duration of 16 Days
  Measurement of safety parameters include physical examinations, clinical laboratory tests, 12-lead ECGs (electrocardiograms) and vital signs.
Number of subjects with adverse events | Up to 30 days
  Total number of subjects with adverse events.
Maximum plasma concentration (Cmax) of the ABT-493 study drug. | (SUB-STUDY 1) Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1. (SUB-STUDY 2) Prior to dosing (0-hour), and at 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period.
  The peak concentration that a drug achieves in a specified compartment after the drug has been administrated and before administration of a second dose.
Area under the plasma concentration-time curve (AUC) for the ABT-493 study drug. | (SUB-STUDY 1) Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1. (SUB-STUDY 2) Prior to dosing (0-hour), and at 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period.
  AUC reflects the actual body exposure to drug after administration of a dose of the drug.
(SUB-STUDY 1) Area under the plasma concentration-time curve (AUC) from time 0 to infinity for the ABT-530 study drug. | Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1.
  The AUC from time 0 to infinity represents the total drug exposure over time.
Maximum plasma concentration (Cmax) of the ABT-530 study drug. | (SUB-STUDY 1) Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1. (SUB-STUDY 2) Prior to dosing (0-hour), 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period.
  The peak concentration that a drug achieves in a specified compartment after the drug has been administrated and before administration of a second dose.
Area under the plasma concentration-time curve (AUC) for the ABT-530 study drug. | (SUB-STUDY 1) Prior to dosing (0-hour), 1, 2, 3, 4, 6, 9, 12, 16, 24, 36, 48, 72, 96 hours and 144 hours after dosing on Study Day 1. (SUB-STUDY 2) Prior to dosing (0-hour), and at 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period.
  AUC reflects the actual body exposure to drug after administration of a dose of the drug.
(SUB-STUDY 2) Area under the plasma concentration-time curve (AUC) during hemodialysis for the ABT-493 study drug. | Prior to dosing (0-hour), and at 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period. Additional samples will be collected at 4, 5, and 6 hours after dosing on Study Day 1 of Period 2 only.
  The AUC during hemodialysis represents the total drug exposure over time.
(SUB-STUDY 2) Area under the plasma concentration-time curve (AUC) during hemodialysis for the ABT-530 study drug. | Prior to dosing (0-hour), and at 1, 2, 3, 9, 12, 16, 24 hours after dosing on Study Day 1 of each Period. Additional samples will be collected at 4, 5 and 6 hours after dosing on Study Day 1 of Period 2 only.
  The AUC during hemodialysis represents the total drug exposure over time.

CONTACTS AND LOCATIONS:
Overall Officials: David Pugatch, MD, Study Director — AbbVie
Locations (3):
- United States (2):
  - Site Reference ID/Investigator# 132890, Miami, Florida
  - Site Reference ID/Investigator# 132889, Orlando, Florida
- Site Reference ID/Investigator# 137332, Grafton, Auckland, New Zealand

REFERENCES:
- [Derived] Kosloski MP, Zhao W, Marbury TC, Preston RA, Collins MG, Pugatch D, Mensa F, Kort J, Liu W. Effects of Renal Impairment and Hemodialysis on the Pharmacokinetics and Safety of the Glecaprevir and Pibrentasvir Combination in Hepatitis C Virus-Negative Subjects. Antimicrob Agents Chemother. 2018 Feb 23;62(3):e01990-17. doi: 10.1128/AAC.01990-17. Print 2018 Mar. PMID 29263061